CLINICAL TRIAL: NCT02137824
Title: A Modified Sinus Floor Elevation Technique - a Pilot Study on 12 Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Kristina Bertl, PD, DMD, MSc, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Maxillary Sinus; Atrophy
MeSH Terms: conditions — Atrophy

ARMS (1):
- sinus floor elevation (Experimental)
  Interventions: Procedure: sinus floor elevation

INTERVENTIONS:
Procedure: sinus floor elevation

SUMMARY:
The aim of the present study is to establish a modified minimally invasive surgical technique for sinus floor augmentation with a residual bone height of 3-6mm.

Hypothesis: The investigators expect that the present surgical technique allows to achieve an adequate implant bed of at least 10mm height after a healing period of 3-5 months. Further the modification of the technique enables a reduced patient stress level.

ELIGIBILITY:
Inclusion Criteria:

* residual bone height of 3-6mm
* residual bone width of >4mm

Exclusion Criteria:

* not treated periodontal disease
* smoker (>5cig/day)
* acute or chronic sinusitis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-05; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Height of augmentation | after 4-5months

CONTACTS AND LOCATIONS:
Locations (1):
- Bernhard Gottlieb School of Dentistry, Medical University of Vienna, Vienna, Austria